CLINICAL TRIAL: NCT00048984
Title: A Groupwide Biology and Banking Study for Ewing Sarcoma
Brief Title: Diagnostic Study of Tumor Characteristics in Patients With Ewing's Sarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AEWS02B1; NCI-2012-02494 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000257115 (Other: Clinical Trials.gov); COG-AEWS02B1 (Other: Children's Oncology Group); NCI-03-C-0216 (Other: NCI); U10CA098543 (NIH); NCT00063271 (obsolete NCT alias); NCT00228774 (obsolete NCT alias)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Localized Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Metastatic Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive, Peripheral

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Paraffin-embedded blocks of tumor tissue or slides of tumor tissue, and blood specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Basic science (biomarker analysis): Patients undergo various specimen collections, including bone marrow aspirate, paraffin-embedded blocks of tumor tissue or slides of tumor tissue, and blood specimens. These specimens are collected before, during, and after any chemotherapy regimens, during follow-up, and at time of recurrence. Translocation studies are performed on specimens to identify fusion genes, specifically EWS-ETS. Serum IGF1 and IFGBP3 levels are determined. Bone marrow is assessed for minimal residual disease using reverse-transcriptase polymerase chain reaction.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Diagnostic trial to study genetic differences in patients who have Ewing's sarcoma. Genetic testing may help predict how cancer will respond to treatment and allow doctors to plan more effective therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop a mechanism to collect and distribute tumor specimens to various investigators, and a system to prioritize and develop quality-control measures for central data reporting of studies undertaken.

II. To determine the prognostic significance of translocation subtype in Ewing sarcoma; to determine the prognostic significance of translocation negative Ewing sarcoma.

III. To determine the prognostic significance of MRD detection in bone marrow specimens by RT-PCR determination of EWS-ETS fusion genes.

IV. To determine whether serum levels of IGF1, IGFBP3 are of significance in the outcome of patients with Ewing sarcoma.

V. To determine whether RNA expression profiles performed on diagnostic specimens will allow for the identification of newer prognostic categories and potentially new molecular targets for treatment in Ewing sarcoma.

VI. To identify new treatment targets for therapy. Further testing of these potential targets will be carried out in hopes of expediting translation of these findings to the clinic.

VII. To establish a bank of Ewing sarcoma xenografts in SCID/Beige mice. VIII. To establish clinical proteomics as a resource for investigations of altered signaling molecules in the pathogenesis of Ewing sarcoma.

OUTLINE: This is a multicenter study.

Patients undergo various specimen collections, including bone marrow aspirate, paraffin-embedded blocks of tumor tissue or slides of tumor tissue, and blood specimens. These specimens are collected before, during, and after any chemotherapy regimens, during follow-up, and at time of recurrence. Translocation studies are performed on specimens to identify fusion genes, specifically EWS-ETS. Serum IGF1 and IFGBP3 levels are determined. Bone marrow is assessed for minimal residual disease using reverse-transcriptase polymerase chain reaction.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or recurrent Ewing's sarcoma
* Availability of the following specimens:

  * Paraffin-embedded block or 20 unstained slides and 1-3 thick (50 micron) sections from initial biopsy
  * Pretreatment serum and whole blood
* Concurrent therapy is not required

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who have Ewing's sarcoma
Sampling Method: Probability Sample
Enrollment: 637 (Actual)
Dates: Start 2003-01; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 1 year
  Univariate analysis using the proportional-hazards regression model will be used to formally assess the prognostic significance of each biological characteristic as it relates to risk for adverse event. Methods such as recursive partitioning adapted to survival analysis will be used to explore possible interactions between the presence of various markers and risk for adverse event.

SECONDARY OUTCOMES:
Success rate in which biomarker analyses can be carried out | Up to 5 years
Percent of the population on which biomarker analysis could be successfully conducted | Up to 5 years
  Determined by the number of patients on whom a definitive analytic result could be obtained, divided by the total number of patients enrolled after the test became part of the routine battery used by the investigators.
Percent of submissions on which biomarker analysis could be successfully conducted | Up to 5 years
  Determined by the number of patients on whom a definitive analytic result could be obtained, divided by the total number of patients for whom a specimen was submitted for the relevant assay.
Relation to known prognostic factors including the presence or absence of metastatic disease, the site of disease, and other known risk factors | Up to 5 years
  The prevalence of these risk factors will be determined for the evaluable and nonevaluable samples to ensure the comparability of these two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel West, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States